CLINICAL TRIAL: NCT03325621
Title: Phase 2a Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Repeated Administrations Over 4 Weeks of the Hepcidin Antagonist PRS-080#022-DP in Anemic Chronic Kidney Disease Patients Undergoing Hemodialysis
Brief Title: Phase 2a Study to Evaluate PRS-080 in Anemic Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pieris Pharmaceuticals GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCS_03_16
Record Dates: First submitted 2017-10-19; First posted 2017-10-30 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2018-11

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: Hepcidin; Hemoglobin; Iron; Anemia of chronic disease

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, placebo-controlled, two dose groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRS-080#022-DP (Active Comparator): Experimental: PRS-080#022-DP Hepcidin antagonist, repeated administrations, ascending doses
  Interventions: Biological: PRS-080#022-DP
- PRS-080-Placebo#001 (Placebo Comparator): Experimental: PRS-080-Placebo#001 Comparator treatment, repeated administrations
  Interventions: Biological: PRS-080-Placebo#001

INTERVENTIONS:
Biological: PRS-080#022-DP — Biological/Vaccine: PRS-080#022-DP Hepcidin antagonism to mobilize iron and to treat anemia
  Other Names: PRS-080
  Arms: PRS-080#022-DP
Biological: PRS-080-Placebo#001 — Placebo Comparator
  Other Names: Placebo
  Arms: PRS-080-Placebo#001

SUMMARY:
Anticalin® proteins are engineered human proteins that are able to bind specific target molecules. The Anticalin PRS-080#022-DP to be investigated in this study is directed against hepcidin and is intended for the treatment of anemia of chronic disease. This pilot Phase 2a study shall investigate the safety, pharmacokinetics and pharmacodynamics of repeated administrations of PRS-080#022-DP in anemic stage 5 chronic kidney disease (CKD) patients undergoing hemodialysis.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled, multiple ascending dose, pilot Phase 2a study in anemic stage 5 chronic kidney disease patients requiring hemodialysis. Eligible patients will undergo screening assessments and PRS-080#22-DP will be administered by intravenous infusion. The study will consist of 2 dose cohorts of 4 mg/kg and 8 mg/kg body weight with 6 patients in each cohort. Using a standard 4+2 design, 4 patients in each cohort will be randomized to PRS-080#022-DP and 2 patients in each cohort will be randomized to placebo. The decision to escalate the dose will be based on an interim analysis of clinical and laboratory safety as well on a comparison with pharmacokinetic data. Safety and tolerability, pharmacokinetics, pharmacodynamics as well as potential immunogenicity will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 5 CKD having been on hemodialysis for at least 90 days;
* Male and post-menopausal (no menses for at least 12 months without an alternative medical cause) female patients with an age of ≥18 years and with a maximum body weight of 85 kg;
* Patients being on stable erythropoiesis stimulating agent dose for 4 weeks prior to Screening;
* Patients being on stable oral or intravenous iron doses for 4 weeks prior to Screening;
* Mean of 3 Hb values during the screening period, each obtained at least 7 days apart must be ≤10.5 g/dL, with a difference of ≤1.0 g/dL between the lowest and highest value;
* Serum ferritin concentration ≥300 ng/mL;
* Transferrin saturation ≤30%;
* Plasma hepcidin concentration at least 5 nmol/L;
* Screening serum folate and vitamin B12 ≥lower limit of normal Hepcidin 5 - 50 nmol/L;
* Male patients with a female partner of childbearing potential agree to use a medically acceptable method of contraception (e.g., condoms, sexual abstinence, vasectomy), not including the rhythm method for 30 days after administration of the study medication; and
* The patient is legally competent, has been informed of the nature, the scope and the relevance of the study, voluntarily agrees to participation and the study's provisions, and has duly signed the informed consent form (ICF). Patient agrees to comply with the protocol-mandated procedures and visits.

Exclusion Criteria:

* Anemia due to causes other than chronic kidney disease, including hemoglobinopathies, hemolytic anemias, myelodysplasia or malignancy;
* Blood transfusion within 2 months before administration of study medication;
* Previous enrollment in this study;
* Patients treated with PRS-080#022-DP in a previous clinical study;
* Current or previous (within 60 days or 5 half-lives before study medication administration) treatment with another investigational drug and/or medical device or participation in another clinical study;
* Employees of the sponsor or patients who are employees or relatives of the investigator;
* Known allergy to any component of the PRS-080#022-DP formulation;
* Positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibody (anti-hepatitis C virus Ab), or human immunodeficiency virus (HIV), serology test results not older than 3 months are accepted;
* Planned surgery during the study period;
* Known or suspected active infection;
* Active or chronic gastrointestinal bleeding, or known coagulation disorder;
* Unwilling or unable to comply with the protocol, in the judgment of the investigator;
* Unstable angina, myocardial infarction, percutaneous transluminal coronary angioplasty/stents, apoplexy (sudden circulatory disturbances of an organ or specific region of the body) or coronary artery bypass grafting <3 months prior to Screening;
* Congestive heart failure: New York Heart Association Class III or IV;
* Peripheral arterial disease with necrosis, stage IV (Fontaine) or grade III (category 5 and 6, Rutherford); and
* Any medical condition that in the judgment of the investigator might interfere with study participation or jeopardize patient's safety during the study (e.g., active infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | 112 days
  Composite measure including signs and symptoms, changes from baseline heart rate and blood pressure, ECG, body temperature, respiratory rate clinical chemistry and hematology

SECONDARY OUTCOMES:
Cmax | 112 days
  Measuring the maximum concentration of PRS-080#022 in the blood
Effects of PRS-080#022 on serum iron | 56 days
  Changes in total serum iron concentration compared to baseline
Effects of PRS-080#022 on ferritin | 56 days
  Changes in serum ferritin concentration compared to baseline
Effects of PRS-080#022 on transferrin saturation | 56 days
  Changes in serum transferrin saturation compared to baseline
Effect of PRS-080#022 on hepcidin concentrations in plasma | 56 days
  Changes in hepcidin concentration compared to baseline
Number of patients developing anti-drug antibodies | 112 days
  Number of patients with antibodies against PRS-080#022 at day 28 compared to baseline
Effects on red blood cell Hb concentration | 56 days
  Changes in Hb concentration compared to baseline
ctrough | 112 days
  Measuring the concentration of PRS-080#022 before the drug application
tmax | 112 days
  Evaluation of the time for PRS-080#022 to reach maximum concentration
Elimination of PRS-080#022 | 112 days
  Evaluation of Terminal rate constant and terminal half-life (t½ ) after the very last administration of PRS-080 in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Renders, Prof. MD, Principal Investigator — Technical University, Munich; Ondřej Viklický, Prof.MD, Principal Investigator — Institute of Clinical and Experimental Medicine Nephrology Clinic Prague
Locations (6):
- Czechia (4):
  - University Hospital Brno, Brno
  - HDS - Klaudian's Hospital, Mladá Boleslav
  - Institute of Clinical and Experimental Medicine (ICEM), Prague
  - VFN Strahov, Prague
- Germany (2):
  - MZV DaVita, Düsseldorf
  - Technical University Munich, Munich

IPD SHARING:
Plan to Share IPD: No